CLINICAL TRIAL: NCT05390762
Title: Evaluation of the Functional Efficacy of a Multidisciplinary Telecare Rehabilitation Program in Chronic Low Back Pain with Psychological Retention and Predominant Sociability : Single Center Randomized Controlled, Single-blind Trial
Brief Title: Telecare Rehabilitation Program in Chronic Low Back Pain with Psychological Retention and Predominant Sociability
Acronym: TELELOMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A00129-34
Record Dates: First submitted 2022-05-06; First posted 2022-05-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluations will be performed by blind operators of the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional care in a day hospital (Active Comparator): 1. A common face to face day hospital, combining physical therapies with psychotherapeutic support such as Cognitive Behavioral Therapy to combat kinesiophobia.
  2. A Second phase of 5 weeks of care face to face day hospital of the reconditioning type of 15 sessions.
  Interventions: Other: Common phase; Other: Care in Face to Face
- Telecare rehabilitation (Experimental): 1. A common face to face day hospital, combining physical therapies with psychotherapeutic support such as Cognitive Behavioral Therapy to combat kinesiophobia.
  2. A Second phase of 5 weeks of Telecare rehabilitation of the reconditioning type of 15 sessions.
  Interventions: Other: Common phase; Other: Telecare rehabilitation

INTERVENTIONS:
Other: Common phase — A common face to face day hospital combining physical therapies with psychotherapeutic support such as Cognitive Behavioral Therapy to combat kinesiophobia.
Other: Telecare rehabilitation — A Second phase of 5 weeks of telecare rehabilitation of the reconditioning type of 15 sessions.
  Arms: Telecare rehabilitation
Other: Care in Face to Face — A Second phase of 5 weeks of care in face to face day hospital of the reconditioning type of 15 sessions.
  Arms: Conventional care in a day hospital

SUMMARY:
The present study proposes to evaluate the impact of a multidisciplinary biopsychosocial Telecare rehabilitation program at the functional level in people with chronic low back pain with major psycho-behavior maintenance. The hypothesis is that a personalized program combining remote psycho-professional and physical care by digital tools improves functional evaluation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (evolution of more than 3 months)
* Patient treated for this pathology in a multidisciplinary program
* Dallas score > 50% in anxiety/depression and sociability dimensions
* Patient who has given free and informed consent to participate in the research
* Patient affiliated to a social security scheme or beneficiary of such a scheme.
* Patient with an internet connection at home, allowing videoconferencing and a digital tool with web cam (tablet or computer).

Exclusion Criteria:

* Recent spine surgery (< 3 months at inclusion visit)
* Cardiovascular risk factor contraindicating sports practice.
* Severe psychiatric pathology
* Low back pain of tumoral or inflammatory origin.
* Associated motor or sensory, neurological impairment.
* Disabling root irradiation
* Pregnant or breastfeeding women
* Patients under legal protection (guardianship, curators or safeguard of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 3 months after the end of rehabilitation
  Overall score of the Oswestry self-questionnaire. The score goes from 0 to 50, It will be converted into a percentage (Score ODI). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Economic efficiency | At the end of the rehabilitation
  The economic efficiency of personalized rehabilitation at the end of the rehabilitation measured by the cost of transport evaluated according to the functional evolution by Oswestry.
Spontaneous pain | At the end of the rehabilitation and 3 month after.
  The spontaneous pain measured by Visual Analogic Scale, from 0 to 100. The 0 represents no pain at all and 100 the worth pain imaginable.
Overall flexibility | At the end of the rehabilitation and 3 month after.
  Measured finger ground distance in centimeters. The patient is asked to touch the ground with both hands while standing with the knees in extension. The distance between the fingertip and the ground is recorded. Higher the distance is, the better it is.
Range of motion of lumbar mobility | At the end of the rehabilitation and 3 month after.
  Active range of motion of lumbar flexion and lumbar extension will be measured with two inclinometers. Higher the score is, the better it is.
Sub pelvis muscle flexibility. | At the end of the rehabilitation and 3 month after.
  The sub pelvis muscle flexibility will be measured by goniometry and centimetry. Higher the score is, the better it is.
Quadriceps strength | At the end of the rehabilitation and 3 month after.
  Testing will be done 90 degrees of knee flexion using a wall. The maximum holding time will be determined with a chronometer (in seconds). Higher the score is, the better it is.
Endurance of trunk extensors | At the end of the rehabilitation and 3 month after.
  Measured by the Sorensen-Biering Test (duration in seconds), higher the score is, the better it is.
Endurance of trunk flexors | At the end of the rehabilitation and 3 month after.
  Measured by the Shirado test (duration in seconds), higher the score is, the better it is.
Anxiety and depression | At the end of the rehabilitation and 3 month after.
  The Anxiety and depression are assessed by the self administered Hospital Anxiety and Depression scale (HAD). It has 14 items from 0 to 3. 7 questions concern, depression and 7 anxiety. The total for each scale is 21. If the score is less than 7, there in no symptomatology.
The kinesiophobia | At the end of the rehabilitation and 3 month after.
  Assessment of the kinesiophobia index by the TAMPA questionnaire. There are 17 questions, from 1 to 4. If the score is high (more than 40 on 68), the kinesiophobia is significant.
Functional abilities | At the end of the rehabilitation and 3 month after.
  Evaluation of the functional disability with the dallas pain questionnaire. It's divided in 4 parts : impact on daily activities, impact on the relation between professional activities and leisure, impact on the relation between anxiety and depression and the impact on sociability. The Dallas questionnaire evaluated the impact of pain from 0 (no impact) to 100% (maximum impact).
Socio professional criteria | 3 months after the end of rehabilitation
  The rate of patients having resumed a professional activity and condition of resumption (part-time therapeutic or not, previous position or adapted position).
Compliance | At the end of the rehabilitation
  Self-assessment compliance evaluated by an adherence booklet
Acceptability | At the end of the rehabilitation program and 3 months after.
  The acceptability will be assessed using a 18-item questionnaire based on the Unified Theory of Acceptance and Use of Technology (UTAUT) model. Each questions are based on a Likert-type 5 point scale ranging from : 1=In total disagreement, 2= Somewhat disagree, 3= Neither agree nor disagree, 4= Somewhat agree, 5=In total agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Jephté Houedakor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pôle Saint-Hélier, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No